CLINICAL TRIAL: NCT05854420
Title: Modified Anterior Lamellar Recession for All Grades of Upper Eyelid Trachomatous Cicatricial Entropion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab Tharwat, Principal Investigator, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Modified ALR
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Entropion
MeSH Terms: conditions — Entropion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified anterior Lamellar Recession (Experimental): All patients in this arm underwent a combination of ALR, blepharoplasty, suprasternal fixation, and cauterization or internal bulb extirpation of posteriorly located lashes.
  Interventions: Procedure: Modified anterior Lamellar Recession

INTERVENTIONS:
Procedure: Modified anterior Lamellar Recession — ALR is one of the procedures used to treat cicatricial entropion and trichiasis. Few studies present the effect of modifications to this procedure in trachomatous entropion and trichiasis. Because trachoma is common in our country, there is a probability that the number of surgeries for TT will rise.

SUMMARY:
This study aims to assess the combination of anterior lamellar recession (ALR) with blepharoplasty, suprasternal fixation, and internal eyelash bulb extirpation of aberrant lashes posteriorly located in patients with any grade of upper eyelid trachomatous cicatricial entropion

ELIGIBILITY:
Inclusion Criteria:

* All patients presented with upper lid trachomatous cicatricial entropion associated with rubbing lashes.
* Patients having a history of argon laser ablation, electrolysis, epilation, or past unsuccessful surgery were also included

Exclusion Criteria:

* Patients with a follow-up period of fewer than 12 months.
* Patients with very severe UCE and required posterior lamellar grafts.
* Patients with etiology other than trachoma.
* Patients with dysplastic lashes without entropion were excluded

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Success rate | 3 months post operative
  The cases will be considered succeed if there is no recurrence of the entropion
Success rate | 6 months post operative
  The cases will be considered succeed if there is no recurrence of the entropion
Success rate | 9 months post operative
  The cases will be considered succeed if there is no recurrence of the entropion
Success rate | 12 months post operative
  The cases will be considered succeed if there is no recurrence of the entropion

CONTACTS AND LOCATIONS:
Locations (1):
- Ehab tharwat, Damietta, New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No